CLINICAL TRIAL: NCT04494945
Title: Approaches to Identify and Care for Individuals With Inherited Cancer Syndromes
Brief Title: Identifying and Caring for Individuals With Inherited Cancer Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jackie Shannon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00020629; NCI-2020-04627 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020629 (Other: OHSU Knight Cancer Institute); U01CA232819 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: BRCA1/2-Associated Hereditary Breast and Ovarian Cancer Syndrome; Breast Ductal Carcinoma In Situ; Hematopoietic and Lymphoid System Neoplasm; Hereditary Neoplastic Syndrome; Lynch Syndrome; Malignant Solid Neoplasm
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Carcinoma, Intraductal, Noninfiltrating; Neoplastic Syndromes, Hereditary; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (genetic testing) (Other): Patients undergo collection of saliva samples for genetic testing. If genetic test is positive, patients receive genetic counseling.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Counseling; Other: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva sample
  Other Names: Biological Sample Collection
Other: Genetic Counseling — Receive genetic counseling if testing results are positive
Other: Genetic Testing — Undergo genetic testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
Other: Survey Administration — Complete a survey

SUMMARY:
This trial examines approaches to identify and care for individuals with inherited cancer syndrome. The purpose of this study is to offer no cost genetic testing to the general public. Researchers hope to learn the value of providing broad, public-wide testing for high risk cancer types (like hereditary breast and ovarian cancer or Lynch syndromes) instead of only testing people whose families are known to be high risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the effectiveness and sustainability of heritable cancer syndrome testing in two proposed screening populations compared to current guidelines.

SECONDARY OBJECTIVES:

I. Measure adherence to current guidelines for screening and prophylactic intervention of Cohorts B and C compared to Cohort A to show non-inferiority.

II. Measure the efficiency of cascade testing (defined as the ratio of family members screened over total possible) for Cohorts B and C compared to Cohort A to show non-inferiority.

III. Determine the costs and effectiveness, specifically quality adjusted life years (QALYs) associated with genetic screening models based on Cohorts B and C to estimate incremental cost-effectiveness ratio (ICER) and show that the costs per QALY are below the acceptable cost effectiveness threshold.

OUTLINE:

Patients undergo collection of saliva samples for genetic testing. If genetic test is positive, patients receive genetic counseling. Patients also complete a survey about cancer prevention, screening, and treatment.

ELIGIBILITY:
Inclusion Criteria:

* ALL COHORTS: 18 years of age or older
* Retrospective COHORT A: Per HIPAA waiver, Retrospective Cohort A will not actively consent
* Retrospective COHORT A: Patients may or may not be diagnosed with cancer
* Retrospective COHORT A: Patients have received genetic counseling in the past 5 years
* Retrospective COHORT A: Patients have genetic variants that include BRCA1, BRCA2 and/or Lynch syndrome
* COHORT A: Per Health Insurance Portability and Accountability Act (HIPAA) waiver, Cohort A returns survey as consent
* COHORT A: Patients may or may not be diagnosed with cancer
* COHORT A: Patients have received genetic counseling in the past 1 - 2 years
* COHORT A: Patients have genetic variants that include BRCA1, BRCA2 and/or Lynch syndrome
* COHORT A: INCLUSIVE of no contact list to exclude from Cohort B
* COHORT B: Creation of secure Healthy Oregon Project (HOP) app account
* COHORT B: Consent to this project, either hard or electronic signature
* COHORT B: Consent to the HOP repository, either hard or electronic signature
* COHORT B: Choosing to submit a deoxyribonucleic acid (DNA) sample
* COHORT B: Patients diagnosed with any National Cancer Institute (NCI)-reportable cancers, including ductal carcinoma in situ (DCIS) and/or in situ breast cancer
* COHORT B: Must have had an encounter within past twelve months
* COHORT B: Exclude Cohort A
* COHORT C: Creation of secure Hop app account
* COHORT C: Consent to this project, either hard or electronic signature
* COHORT C: Consent to the HOP repository, either hard or electronic signature
* COHORT C: Choosing to submit a DNA sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27500 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and sustainability of heritable cancer syndrome testing in the two novel testing populations | Up to 5 years
  Determine the costs and effectiveness, specifically Quality Adjusted Life Years (QALYs) associated with genetic screening models based on Cohorts B and C to estimate incremental cost-effectiveness ratio (ICER) and show that the costs per QALY are below the acceptable cost effectiveness threshold.
Adherence to standard of care for hereditary breast and ovarian cancer (HBOC) and Lynch syndromes | Up to 5 years
  For Lynch syndrome we identify compliance as colonoscopy in past two years and bilateral salpingo-oophorectomy (BSO ) after child-bearing age. For HBOC, compliance is defined as breast imaging in past year or risk reducing surgery at any point in women.
Merged risk reduction strategies of bilateral salpingo-oophorectomy (BSO) or bilateral mastectomy and imaging | Up to 5 years
  The merged risk reduction strategies of BSO or bilateral mastectomy and the imaging are treated as evidence of risk reducing behavior.
Cascade screening rate among Lynch or HBOC positive carriers | Up to 5 years
  Will conduct negative binomial regression model and non-inferiority will be determined by rate ratio and its 95% confidence interval (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Jackilen Shannon, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - Providence Portland Medical Center, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Data and samples collected under this protocol will be stored indefinitely in this study's repository for future research use. Participants must agree to future research use of their samples/data to participate in HOP.
  Data/samples from participants who identify as American Indian/Alaska Native will be flagged within the HOP database so they can be excluded from data/sample releases for research purposes.
  HOP has created a Data Access Committee (DAC) to review all requests for HOP data/samples. The DAC will review requests for feasibility and scientific merit before any data/samples are released.
  OHSU investigators wishing to receive data from this study will sign a data release agreement documenting they will:
  * Meet all IRB requirements (IRB approval, exemption or nonhuman subjects research determination), as appropriate.
  * Use data only for the research described in their data request and/or IRB application/ protocol and obtain additional IRB approval if secondary studies are